CLINICAL TRIAL: NCT04106336
Title: Cortical Excitability and Role of rTMS in Cannabis Use Disorder
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Omar Radwan Helal, Asmaa Omar Radwan Helal, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rTMS in cannabis use disorder
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cannabis Use Disorder, Moderate
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non cannabis addict (No Intervention): 30 non cannabis addict will be control group
- cannabis addict (Active Comparator): 30 cannabis addict will undergo rTMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Repetitive transcranial magnetic stimulation (rTMS) will be done for cannabis addict
  Arms: cannabis addict

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) and cortical excitability have a role in cannabis use disorder

ELIGIBILITY:
Inclusion Criteria:

* 18to 50 years of age
* cannabis use disorder according to DSM 5 definition
* clear consent to participate in study

Exclusion Criteria:

* cardiac peacemaker
* metal implant in the head as participate will be applied to magnetic field of TMS
* current intake of any medication affect cognition (as anti psychotic and anti epileptic)
* current history of neurological , psychiatric or general medical disease .current or previous drug (other than cannabis )or alcohol abuse or participation in another trial during the past 8 weeks .
* age younger than 18 and older than 50 years

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Determination of role of rTMS for reducing cannabis craving | 1 year
  Incidenc of cannabis craving after rTMS

SECONDARY OUTCOMES:
Estimation of cortical excitability in cannabis addict | 1 year
  Incidence of cannabis craving after cortical excitability